CLINICAL TRIAL: NCT06882915
Title: Efficacy and Safety of Trifluridine/tipiracil (TAS-102) Combined with Bevacizumab and Putalimab in the Treatment of Patients with MCRC After Cytoreductive Surgery: a Single-arm, Single-center Clinical Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0383
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: The treatment regimen is trifluridine/tipirimidine (TAS-102) combined with bevacizumab and putelimab, with a 28-day medication cycle.
  TAS-102: Use at the recommended dose of 35 mg/m² each time, twice a day from the 1st to the 5th day and the 8th to the 12th day every 28 days, with meals.
  Bevacizumab: Once a day on the 1st and 15th day every 28 days, at the recommended dose of 5 mg/kg each time, with meals.
  Putelimab: According to the recommended dose of 200 mg/time, intravenous drip, infusion time is 60 minutes, once every 28 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trifluridine/tipiracil (TAS-102) combined with bevacizumab and ptemizumab (Experimental): TAS-102: Use at the recommended dose of 35 mg/m² each time, twice a day on the 1st to 5th day and the 8th to 12th day every 28 days, with meals.
  Bevacizumab: Once a day on the 1st and 15th day every 28 days, at the recommended dose of 5 mg/kg each time, with meals.
  Putlimumab: At the recommended dose of 200 mg/time, intravenous drip, infusion time is 60 minutes, once every 28 days.
  Interventions: Drug: Trifluridine/tipiracil (TAS-102) combined with bevacizumab and ptemizumab

INTERVENTIONS:
Drug: Trifluridine/tipiracil (TAS-102) combined with bevacizumab and ptemizumab — TAS-102: Use at the recommended dose of 35 mg/m² each time, twice a day on the 1st to 5th day and the 8th to 12th day every 28 days, with meals.
  Bevacizumab: Once a day on the 1st and 15th day every 28 days, at the recommended dose of 5 mg/kg each time, with meals.
  Putlimumab: At the recommended dose of 200 mg/time, intravenous drip, infusion time is 60 minutes, once every 28 days.

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignant tumors. With the rapid development of China's economy, people's living standards have been significantly improved, and lifestyles and dietary structures have changed. Smoking, drinking, high-fat, high-energy diets, etc. have led to an increase in the incidence of colorectal cancer year by year. Data show that in 2022, there will be 510,000 new cases of colorectal cancer in China, and about 240,000 deaths related to colorectal cancer. Radical surgery is the main initial treatment for early and middle-stage colorectal cancer and some metastatic colorectal cancer. Although the level of surgical treatment of colorectal cancer has been greatly improved and can achieve cure for some patients, its 5-year overall survival rate is only about 60%, and the main cause of death is distant metastasis and recurrence. In recent years, with the in-depth understanding of the treatment mechanism of metastatic colorectal cancer (mCRC), a variety of new treatment options have been proposed and applied in clinical practice in order to improve the quality of life of patients and prolong their survival.

Trifluridine/tipivirine (TAS-102) is a new type of cytotoxic drug that exerts anti-tumor effects by directly incorporating into DNA chains to destroy DNA function. Its mechanism of action is different from that of fluorouracil drugs, and it can resist 5-fluorouracil (5-FU) resistance, providing a new treatment option for mCRC patients. TAS-102 has been approved in China for mCRC patients who have previously received fluoropyrimidine, oxaliplatin, and irinotecan-based chemotherapy, as well as those who have previously received or are not suitable for anti-vascular endothelial growth factor (VEGF) therapy and anti-epidermal growth factor receptor (EGFR) therapy (RAS wild type). Bevacizumab, as a monoclonal antibody targeting VEGF, exerts its anti-tumor effect by inhibiting tumor angiogenesis. Putlimumab, as an immune checkpoint inhibitor, enhances the body's immune response to tumors by blocking the PD-1/PD-L1 signaling pathway.

Combination therapy has attracted much attention due to its possible synergistic effect. Studies have shown that TAS-102 combined with bevacizumab can achieve longer overall survival (OS) than TAS-102 monotherapy. In addition, TAS-102 combined with bevacizumab for refractory mCRC has also been approved by the FDA, showing its potential and importance in the treatment of mCRC. Therefore, this study aims to explore the efficacy and safety of TAS-102 combined with bevacizumab and putelimab in patients with mCRC after cytoreductive surgery, in order to provide a more effective treatment for mCRC patients. Through the design of a single-arm, single-center clinical study, we can have a deeper understanding of the efficacy and safety of this combined treatment in a specific patient population, providing a scientific basis for future clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* 1. After complete cytoreduction surgery (CC0) for peritoneal metastasis of colorectal cancer;
* 2. Patients diagnosed with peritoneal metastasis of colorectal cancer by pathology and imaging;
* 3. Microsatellite stable (MSS) by genetic testing;
* 4. Expected survival time at least 6 months;
* 5. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1;
* 6. Normal function of the heart, liver and kidneys;
* 7. Normal hematological indicators: neutrophil count ≥1.5×109/L, white blood cell count (WBC) ≥3.0×109/L, hemoglobin ≥10g/dL, platelet count ≥100×109/L;
* 8. Normal biochemical indicators: total bilirubin ≤1.5×upper limit of normal (ULN), AST and ALT ≤2.5 times upper limit of normal, serum creatinine and urea nitrogen (BUN) ≤1.5 times the upper limit of normal value;

Exclusion Criteria:

* 1. Unwilling to sign the informed consent form;
* 2. Currently participating in interventional research treatment, or receiving other drugs or research devices within 4 weeks before enrollment;
* 3. Having other malignant tumors at the same time;
* 4. Other serious diseases that the investigators judge may affect follow-up and short-term survival;
* 5. Allergic to TAS-102, bevacizumab or putelimab components;
* 6. Uncontrolled brain metastases;
* 7. Pregnant or lactating women;
* 8. Those with a history of mental illness;
* 9. Uncontrolled complications including but not limited to active infection, symptomatic congestive heart failure, unstable angina, arrhythmia;
* 10. Severe coronary artery disease or cerebrovascular disease, or other diseases that the investigators believe are not suitable for enrollment;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Two Years
  The period from the beginning of treatment to the first occurrence of disease progression or death from any cause. If such situation is not met, the last evaluation date shall be used for analysis. In addition, if the treatment is terminated without confirming the progress of the disease, the imaging examination and follow-up should also be carried out after the treatment is terminated.

SECONDARY OUTCOMES:
Objective Remission Rate (ORR) | Two Years
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit. The remission period usually refers to the period from the beginning of curative effect to the confirmation of tumor progression. The objective response rate is generally defined as the sum of complete response plus partial response (CR+PR).
Overall Survival (OS) | Two Years
  The time from the date of treatment to the date of death due to any reason. For patients who survived in the final analysis, the date of the last contact will be recorded.
Treatment response | Two Years
  To evaluate tumor response using imaging examinations (CT/MRI) and tumor shrinkage rate using the response evaluation criteria in solid tumors (RECIST 1.1).
Incidence rate of adverse events | Baseline before any treatment,3 months after any treatment
  According to NCI CTCAE v5.0